CLINICAL TRIAL: NCT04201548
Title: Comparison of Clinical and Physiological Response Among Three Modalities of Exercise Training in COPD With Chronic Respiratory Failure (CRF)
Brief Title: Different Modalities of Exercise Training in COPD With Chronic Respiratory Failure (CRF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: Universita di Verona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE2288
Record Dates: First submitted 2019-11-28; First posted 2019-12-17 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Copd; Chronic Hypoxemic Respiratory Failure
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Endurance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active Comparator (Active Comparator): This is the constant-load Endurance Training (ET) group which will constitute the control group.
  Interventions: Other: Endurance Training
- Long High Intensity Interval Training (Experimental): This is the Long High Intensity Interval Training (Long-HIIT) group.
  Interventions: Other: Long High Intensity Interval Training
- Short High Intensity Interval Training (Experimental): This is the Short High Intensity Interval Training (Short-HIIT) group.
  Interventions: Other: Short High Intensity Interval Training

INTERVENTIONS:
Other: Endurance Training — These patients will perform an aerobic exercise with a moderate intensity cycle ergometer. The exercise session on an exercise bike will last 33 minutes at a constant load, starting from an intensity equal to the load of 60% of the maximum load (max watt) achieved at the incremental test.
  Working volume = 60 X 33 = 1980
  Other Names: ET; Active Comparator
  Arms: Active Comparator
Other: Long High Intensity Interval Training — The patients assigned to the Long-HIIT group will perform a 32-minute interval work with 4x4 protocol (active phase x passive phase) performing 4 minutes at an intensity of 80-85% of the Max Watt (active phase) spaced from 4 minutes to 40% of the Max Watt (passive phase). The goal of high intensity work will be to bring the heart rate to a level close to 85-90% of the maximum cardiac frequency achieved in the incremental exercise test. If this target is not reached within the session, the load of the next one will be increased in the following session with 10 watt steps.
  Working volume = 16 X 85 + 16 x 40 = 2000
  Other Names: Long-HIIT; Experimental 1
  Arms: Long High Intensity Interval Training
Other: Short High Intensity Interval Training — The patients assigned to the Short-HIIT group will perform an interval work with initial intensity equal to 100% of the Max Watt highlighted in the incremental exercise stress test in the phase (30 seconds) followed by a passive phase of 30 seconds at 50% of the Max Watt for a period of 26 minutes a day. The intensity will be gradually increased during the sessions with symptom-based progression, according to the protocol of Maltais et al. with steps of 10 watts each increment.
  Working volume = 13 X 100 + 13 x 50 = 2050
  Other Names: Short-HIIT; Experimental 2
  Arms: Short High Intensity Interval Training

SUMMARY:
Advanced Chronic Obstructive Pulmonary Disease (COPD) is a condition with a negative prognosis that causes symptoms such as wheezing and fatigue that dramatically reduce the quality of life of the person with the disease.

Typically, the advanced stage of COPD is characterized by a fluctuating pattern and recurrent hospitalizations, and by a vicious circle in which dyspnoea increases and exercise tolerance reduces, causing depression with social isolation, low quality of life and increased risk of death.

Muscle dysfunction in these patients contributes together with dynamic hyperinflation to increased fatigue and dyspnoea during exercise, leading to early interruption of exertion, before reaching the maximal aerobic capacity.

The European and American guidelines of the American Thoracic Society / European Respiratory Society relating to the patient with COPD emphasize the need for the patient to undergo Respiratory Rehabilitation (RR) programs. The RR should include training programs as they improve exercise capacity, dyspnoea and quality of life more than programs that do not include training.

To our knowledge, no study has been performed in COPD with chronic respiratory failure (CRF) patients to evaluate the effects of High Interval Training compared to continuous submaximal training. Moreover, no different interval training protocols have been compared. However, studies conducted on healthy subjects or on other pathologies, show how the interval training protocol induces, in a specific and diversified way, physiological modifications to the cardio-respiratory and muscular systems.

In COPD patients with respiratory failure with marked muscular dysfunction and associated systemic changes (systemic inflammation, vascular changes, pulmonary hypertension, right heart failure, etc.), the evaluation of the best training program would reinforce the rehabilitative indications not yet fully proposed in the Guidelines. Moreover, the evaluation of the response to different training stimuli could provide important information on the reversibility of the intolerance to the effort in this patient population.

Primary aim of this study will be to evaluate the physiological effects on exercise tolerance of three training modalities performed in an intra-hospital setting (classic endurance training compared to two high-intensity interval programs - Long Interval Training and Short Interval training) in a population of COPD patients with chronic hypoxemic respiratory failure.

DETAILED DESCRIPTION:
Advanced (Chronic Obstructive Pulmonary Disease) COPD is a condition with a negative prognosis that causes symptoms such as wheezing and fatigue that dramatically reduce the quality of life of the person with the disease.

Typically, the advanced stage of COPD is characterized by a fluctuating pattern and recurrent hospitalizations, and by a vicious circle in which dyspnoea increases and exercise tolerance reduces, which in turn causes depression and associated social isolation, low quality of life and increased risk of death.

Muscle dysfunction in these patients contributes together with dynamic hyperinflation to increased fatigue and dyspnoea during exercise, leading to early interruption of exertion, before reaching maximum aerobic capacity.

The European and American guidelines of the American Thoracic Society / European Respiratory Society relating to the patient with Chronic Obstructive Pulmonary Disease (COPD) emphasize the need for the patient to undergo Respiratory Rehabilitation (RR) programs. The RR should include training programs as they improve exercise capacity, dyspnoea and quality of life more than programs that do not include training.

However, although there are many studies referring to the benefits of physical exercise in patients with COPD with mild-to-moderate severity, the recent guidelines provide few recommendations for types of training and its efficacy for patients with advanced disease that have already developed Chronic Respiratory Failure (CRF) and use of Long Term Oxygen Therapy (LTOT).

Thanks to a retrospective study on 1047 patients, the Authors have previously shown that patients with COPD with CRF respond to a rehabilitation program (in terms of exercise tolerance, blood gases, dyspnoea and quality of life) as well as COPD patients without CRF.

A recent meta-analysis conducted by Paneroni et al. supports the effectiveness of exercise in improving quality of life and functional capacity in patients with severe COPD (FEV1 <35%), with or without CRF. The study showed that so far the training proposed to these patients is mainly of moderate-intensity endurance and performed primarily through the continuous use of exercise bikes or free walking. In a similar way to patients with moderate or mild severity, the setting of the exercise was mainly proposed using a speed or a load that approximates around 70% of the maximum value reached in an incremental test.

Regarding the type of exercise to be used in patients with COPD, several recent papers suggest the opportunity to use interval training even in high intensity. The purpose of the High Interval Training is to repeatedly stress the cardio-respiratory and muscular system, above "what is normally required for normal activities, through" bouts of high intensity and short duration exercise".

In subjects with COPD, this type of training could guarantee a delay in the development of the dynamic hyperinflation mechanism typical of the pathology and could guarantee greater physiological modifications regarding the classical submaximal continuous training. Despite some physiological studies that have tested this effect, the results of the clinical application of these interventions appear - in subjects with moderate COPD - similar to that got with continuing training. However, the protocols proposed to date appear to be diversified in terms of approach, especially concerning the intensity and duration of the active and passive phases.

To our knowledge, no study has been performed in COPD with CRF patients to evaluate the effects of High Interval Training compared to continuous submaximal training and no protocols on different interval training have been compared. Indeed, studies conducted on healthy subjects or on other pathologies, show how the interval training protocol induces, in a specific and diversified way, physiological modifications to the cardiorespiratory and muscular systems.

In patients with respiratory failure with marked muscular dysfunction and associated systemic changes (systemic inflammation, vascular changes, pulmonary hypertension, right heart failure, etc.), the evaluation of the best training program would reinforce the rehabilitative indications not yet fully proposed in the Guidelines. Moreover, the evaluation of the response to different training stimuli could provide important information on the reversibility of the intolerance to the effort in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* age> 50 years
* clinical definition of COPD according to GOLD guidelines (10) with FEV1 / FVC G 70% and FEV1 <50% of the above
* PaO2 in air-ambient lower than 60 mmHg evaluated through arterial blood gas analysis
* oxygen therapy prescription for more than 18 hours/ day for at least one month
* clinical stable condition

Exclusion Criteria:

* presence of pulmonary diseases other than COPD
* respiratory tract infections in the last 4 weeks
* termination

Min Age: 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in effort tolerance | at baseline, 1 month and 7 months
  We will evaluate the time to exhaustion (Tlim) of a Constant Load Endurance Test (CLET) taht will be set at load corresponding to 80% of the Watts max achieved at the incremental cicloergometer test.
Changes in the maximal work load | at baseline and 1 month
  Another way to evaluate changes in effort tolerance will be to evaluate the maximal work load (Watts max) that patients will achive during a cicloergometer incremental test.
Changes in walking distance | at baseline, 1 month and 7 months
  Another way to evaluate changes in effort tolerance will be to evaluate meters walked during a 6 minute walking test (6MWT).

SECONDARY OUTCOMES:
Percentage of drop out patients | at 1 month
  To evaluate feasibility of the study, we will calculate the percentage of patients dropped out at the end of the rehabilitation period
Patient's satisfaction: Likert scale | at 1 month
  To evaluate feasibility of the study, we will administer to patients a questionnaire of satisfaction at the end of the rehabilitation period. Likert scale will be from 0 to 4, where 0= completely unsatisfied and 4= very satisfied)
Change in dyspnoea | at baseline, 1 month and 7 months
  We will evaluated dyspnea by Barthel index Dyspnea, a scale measuring dyspnea during basal activities of daily living (ADL). It is a 10-item scale ranging from 0= absence of dyspnea to 100= maximal dyspnea)
Changes in quadriceps volume | at baseline, 1 month and 7 months
  We will evaluate changes in muscle volume (quadricips) by ecography
Change in ADL performance | at baseline, 1 month and 7 months
  We will evaluate the activities of daily life through the Glittre-ADL test. This consists in a circuit of 5-serie of activities (lifting a chair, walking, lifting 2 steps, moving the weight up and down from a shelf). We will evaluate the total time spent to complete the performance.
Change in fatigue (physiological evaluation) | at baseline, 1 month and 7 months
  We will evaluate the change in force generated by a Maximal Volontary Contraction (MVC) and an Electrically stimulated muscular contractions at rest [Resting Twitch (RT)] of the quadriceps muscle (Q) after a fatiguing task ( CLET). Subjects will be seated upright with a back support. The hip and knee will be flexed at 90 ° and the force will be measured by a force transducer.
  Electromyographic evaluation: the M waves will be recorded by the Q muscle (vastus lateralis). The EMG signals will be amplified with a bandwidth of 10 Hz-1 kHz and digitized online at a sampling frequency of 5 kHz. Voluntary electromyographic activation of the quadriceps muscle during MVC will be evaluated using a superimposed contraction technique.
Change in fatigue (qualitative evaluation) | at baseline, 1 month and 7 months
  For the qualitative evaluation, we will use the Fatigue severity scale that is a 9-item scale ranging from 7= absence of fatigue to 63= maximal presence of fatigue).
Change in Endothelial function | at baseline, 1 month and 7 months
  The endothelial function will be evaluated by an ultrasound evaluation of the common femoral artery before and after the application of the short Passive Leg Movement (sPLM) technique.
Change in Balance | at 1 month and 7 months
  To evaluate balance and consequent risk of falls, a Berg scale will be used. Berg scale is composed by 14 balance related tasks, ranging from score 0=worse balance to 56= best balance.
Change in quality of life | 1 month and 7 months
  COPD Assessment Test (CAT) scale will be used. CAT is a 8-item scale, ranging from score 0 to 40 (where 0=best and 40=worse) evaluating quality of life and well-being
Change in quality of life | at 1 month and 7 months
  MRF scale will be used. MRF is a 28-item questionnaire to assess health outcomes in Chronic Respiratory Failure (CRF). MRF ranges from 26=worse to best = 0
  ...

CONTACTS AND LOCATIONS:
Overall Officials: Mara Paneroni, MSc, PT, Principal Investigator — Istituti Clinici Scientifici Maugeri
Locations (1):
- ICS Maugeri IRCCS, Respiratory Rehabilitation of the Institute of Lumezzane, Lumezzane, Brescia, Italy

REFERENCES:
- [Background] Mirza S, Clay RD, Koslow MA, Scanlon PD. COPD Guidelines: A Review of the 2018 GOLD Report. Mayo Clin Proc. 2018 Oct;93(10):1488-1502. doi: 10.1016/j.mayocp.2018.05.026. PMID 30286833
- [Background] Charususin N, Dacha S, Gosselink R, Decramer M, Von Leupoldt A, Reijnders T, Louvaris Z, Langer D. Respiratory muscle function and exercise limitation in patients with chronic obstructive pulmonary disease: a review. Expert Rev Respir Med. 2018 Jan;12(1):67-79. doi: 10.1080/17476348.2018.1398084. Epub 2017 Nov 6. PMID 29072087
- [Background] Spruit MA, Singh SJ, Garvey C, ZuWallack R, Nici L, Rochester C, Hill K, Holland AE, Lareau SC, Man WD, Pitta F, Sewell L, Raskin J, Bourbeau J, Crouch R, Franssen FM, Casaburi R, Vercoulen JH, Vogiatzis I, Gosselink R, Clini EM, Effing TW, Maltais F, van der Palen J, Troosters T, Janssen DJ, Collins E, Garcia-Aymerich J, Brooks D, Fahy BF, Puhan MA, Hoogendoorn M, Garrod R, Schols AM, Carlin B, Benzo R, Meek P, Morgan M, Rutten-van Molken MP, Ries AL, Make B, Goldstein RS, Dowson CA, Brozek JL, Donner CF, Wouters EF; ATS/ERS Task Force on Pulmonary Rehabilitation. An official American Thoracic Society/European Respiratory Society statement: key concepts and advances in pulmonary rehabilitation. Am J Respir Crit Care Med. 2013 Oct 15;188(8):e13-64. doi: 10.1164/rccm.201309-1634ST. PMID 24127811
- [Background] Carone M, Patessio A, Ambrosino N, Baiardi P, Balbi B, Balzano G, Cuomo V, Donner CF, Fracchia C, Nava S, Neri M, Pozzi E, Vitacca M, Spanevello A. Efficacy of pulmonary rehabilitation in chronic respiratory failure (CRF) due to chronic obstructive pulmonary disease (COPD): The Maugeri Study. Respir Med. 2007 Dec;101(12):2447-53. doi: 10.1016/j.rmed.2007.07.016. Epub 2007 Aug 28. PMID 17728121
- [Background] Paneroni M, Simonelli C, Vitacca M, Ambrosino N. Aerobic Exercise Training in Very Severe Chronic Obstructive Pulmonary Disease: A Systematic Review and Meta-Analysis. Am J Phys Med Rehabil. 2017 Aug;96(8):541-548. doi: 10.1097/PHM.0000000000000667. PMID 28099192
- [Background] Sabapathy S, Kingsley RA, Schneider DA, Adams L, Morris NR. Continuous and intermittent exercise responses in individuals with chronic obstructive pulmonary disease. Thorax. 2004 Dec;59(12):1026-31. doi: 10.1136/thx.2004.026617. PMID 15563700
- [Background] Beauchamp MK, Nonoyama M, Goldstein RS, Hill K, Dolmage TE, Mathur S, Brooks D. Interval versus continuous training in individuals with chronic obstructive pulmonary disease--a systematic review. Thorax. 2010 Feb;65(2):157-64. doi: 10.1136/thx.2009.123000. Epub 2009 Dec 8. PMID 19996334
- [Background] Buchheit M, Laursen PB. High-intensity interval training, solutions to the programming puzzle: Part I: cardiopulmonary emphasis. Sports Med. 2013 May;43(5):313-38. doi: 10.1007/s40279-013-0029-x. PMID 23539308
- [Background] Choudhury G, Rabinovich R, MacNee W. Comorbidities and systemic effects of chronic obstructive pulmonary disease. Clin Chest Med. 2014 Mar;35(1):101-30. doi: 10.1016/j.ccm.2013.10.007. PMID 24507840
- [Background] Norman G. Likert scales, levels of measurement and the "laws" of statistics. Adv Health Sci Educ Theory Pract. 2010 Dec;15(5):625-32. doi: 10.1007/s10459-010-9222-y. Epub 2010 Feb 10. PMID 20146096
- [Background] Vogelmeier CF, Criner GJ, Martinez FJ, Anzueto A, Barnes PJ, Bourbeau J, Celli BR, Chen R, Decramer M, Fabbri LM, Frith P, Halpin DM, Lopez Varela MV, Nishimura M, Roche N, Rodriguez-Roisin R, Sin DD, Singh D, Stockley R, Vestbo J, Wedzicha JA, Agusti A. Global Strategy for the Diagnosis, Management, and Prevention of Chronic Obstructive Lung Disease 2017 Report: GOLD Executive Summary. Arch Bronconeumol. 2017 Mar;53(3):128-149. doi: 10.1016/j.arbres.2017.02.001. Epub 2017 Mar 6. English, Spanish. PMID 28274597
- [Background] American Thoracic Society; American College of Chest Physicians. ATS/ACCP Statement on cardiopulmonary exercise testing. Am J Respir Crit Care Med. 2003 Jan 15;167(2):211-77. doi: 10.1164/rccm.167.2.211. No abstract available. PMID 12524257
- [Background] Holland AE, Spruit MA, Troosters T, Puhan MA, Pepin V, Saey D, McCormack MC, Carlin BW, Sciurba FC, Pitta F, Wanger J, MacIntyre N, Kaminsky DA, Culver BH, Revill SM, Hernandes NA, Andrianopoulos V, Camillo CA, Mitchell KE, Lee AL, Hill CJ, Singh SJ. An official European Respiratory Society/American Thoracic Society technical standard: field walking tests in chronic respiratory disease. Eur Respir J. 2014 Dec;44(6):1428-46. doi: 10.1183/09031936.00150314. Epub 2014 Oct 30. PMID 25359355
- [Background] Parshall MB, Schwartzstein RM, Adams L, Banzett RB, Manning HL, Bourbeau J, Calverley PM, Gift AG, Harver A, Lareau SC, Mahler DA, Meek PM, O'Donnell DE; American Thoracic Society Committee on Dyspnea. An official American Thoracic Society statement: update on the mechanisms, assessment, and management of dyspnea. Am J Respir Crit Care Med. 2012 Feb 15;185(4):435-52. doi: 10.1164/rccm.201111-2042ST. PMID 22336677
- [Background] Gulart AA, Araujo CLP, Munari AB, Santos KD, Karloh M, Foscarini BG, Dal Lago P, Mayer AF. The minimal important difference for Glittre-ADL test in patients with chronic obstructive pulmonary disease. Braz J Phys Ther. 2020 Jan-Feb;24(1):54-60. doi: 10.1016/j.bjpt.2018.11.009. Epub 2018 Nov 20. PMID 30497829
- [Background] Amann M, Romer LM, Subudhi AW, Pegelow DF, Dempsey JA. Severity of arterial hypoxaemia affects the relative contributions of peripheral muscle fatigue to exercise performance in healthy humans. J Physiol. 2007 May 15;581(Pt 1):389-403. doi: 10.1113/jphysiol.2007.129700. Epub 2007 Feb 22. PMID 17317739
- [Background] Broxterman RM, Trinity JD, Gifford JR, Kwon OS, Kithas AC, Hydren JR, Nelson AD, Morgan DE, Jessop JE, Bledsoe AD, Richardson RS. Single passive leg movement assessment of vascular function: contribution of nitric oxide. J Appl Physiol (1985). 2017 Dec 1;123(6):1468-1476. doi: 10.1152/japplphysiol.00533.2017. Epub 2017 Aug 31. PMID 28860173
- [Background] Adami A, Rossiter HB. Principles, insights, and potential pitfalls of the noninvasive determination of muscle oxidative capacity by near-infrared spectroscopy. J Appl Physiol (1985). 2018 Jan 1;124(1):245-248. doi: 10.1152/japplphysiol.00445.2017. Epub 2017 Jul 6. No abstract available. PMID 28684592
- [Background] Gonzalez-Alonso J, Richardson RS, Saltin B. Exercising skeletal muscle blood flow in humans responds to reduction in arterial oxyhaemoglobin, but not to altered free oxygen. J Physiol. 2001 Jan 15;530(Pt 2):331-41. doi: 10.1111/j.1469-7793.2001.0331l.x. PMID 11208980
- [Background] Ryan TE, Brophy P, Lin CT, Hickner RC, Neufer PD. Assessment of in vivo skeletal muscle mitochondrial respiratory capacity in humans by near-infrared spectroscopy: a comparison with in situ measurements. J Physiol. 2014 Aug 1;592(15):3231-41. doi: 10.1113/jphysiol.2014.274456. Epub 2014 Jun 20. PMID 24951618
- [Background] Ryan TE, Southern WM, Reynolds MA, McCully KK. A cross-validation of near-infrared spectroscopy measurements of skeletal muscle oxidative capacity with phosphorus magnetic resonance spectroscopy. J Appl Physiol (1985). 2013 Dec;115(12):1757-66. doi: 10.1152/japplphysiol.00835.2013. Epub 2013 Oct 17. PMID 24136110
- [Background] Sibley KM, Howe T, Lamb SE, Lord SR, Maki BE, Rose DJ, Scott V, Stathokostas L, Straus SE, Jaglal SB. Recommendations for a core outcome set for measuring standing balance in adult populations: a consensus-based approach. PLoS One. 2015 Mar 13;10(3):e0120568. doi: 10.1371/journal.pone.0120568. eCollection 2015. PMID 25768435
- [Background] Jones PW, Harding G, Berry P, Wiklund I, Chen WH, Kline Leidy N. Development and first validation of the COPD Assessment Test. Eur Respir J. 2009 Sep;34(3):648-54. doi: 10.1183/09031936.00102509. PMID 19720809
- [Background] Vidotto G, Carone M, Jones PW, Salini S, Bertolotti G; Quess Group. Maugeri Respiratory Failure questionnaire reduced form: a method for improving the questionnaire using the Rasch model. Disabil Rehabil. 2007 Jul 15;29(13):991-8. doi: 10.1080/09638280600926678. PMID 17612984
- [Background] Helgerud J, Bjorgen S, Karlsen T, Husby VS, Steinshamn S, Richardson RS, Hoff J. Hyperoxic interval training in chronic obstructive pulmonary disease patients with oxygen desaturation at peak exercise. Scand J Med Sci Sports. 2010 Feb;20(1):e170-6. doi: 10.1111/j.1600-0838.2009.00937.x. Epub 2009 May 26. PMID 19793218
- [Background] Vogiatzis I, Terzis G, Nanas S, Stratakos G, Simoes DC, Georgiadou O, Zakynthinos S, Roussos C. Skeletal muscle adaptations to interval training in patients with advanced COPD. Chest. 2005 Dec;128(6):3838-45. doi: 10.1378/chest.128.6.3838. PMID 16354852
- [Background] Maltais F, LeBlanc P, Jobin J, Berube C, Bruneau J, Carrier L, Breton MJ, Falardeau G, Belleau R. Intensity of training and physiologic adaptation in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 1997 Feb;155(2):555-61. doi: 10.1164/ajrccm.155.2.9032194.
- [Result] Paneroni M, Cavicchia A, Beatrice S, Bertacchini L, Venturelli M, Vitacca M. The Influence of Lung Function and Respiratory Muscle Strength on Quadriceps Muscle Fatigability in COPD Patients Under Long-term Oxygen Therapy. Arch Bronconeumol. 2024 Jul;60(7):410-416. doi: 10.1016/j.arbres.2024.04.004. Epub 2024 Apr 23. English, Spanish. PMID 38719676